CLINICAL TRIAL: NCT00277433
Title: Histamine Pharmacogenetics in Children With Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: American College of Clinical Pharmacy (Other); PPRU (Unknown); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: PPRU 10744; 1U10HD045934-01 (NIH)
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Dermatitis, Atopic
Keywords: Atopic Dermatitis; Eczema; Genetics; Histamine
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — buccal-derived DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Atopic Dermatitis
  Interventions: Other: Buccal Swab
- Non-atopic control
  Interventions: Other: Buccal Swab

INTERVENTIONS:
Other: Buccal Swab — collection of buccal swab

SUMMARY:
The primary goal of the study is to investigate the impact of a common genetic polymorphism in a histamine detoxification enzyme that may well have a common role in regulating the expression of atopic dermatitis (AD) and other related atopic diseases in children.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a common condition in the pediatric population, affecting an estimated 15% of all children greater than 18 months of age in the United States. It is now recognized that AD is a disease of significant heterogeneity with respect to both disease severity and response to conventional pharmacologic therapies. With the recognition of this variability comes the understanding that, as with many other allergic disease, there exist many specific disease phenotypes that ultimately govern response to pharmacologic intervention. The characterization of these unique phenotypes and their associated biologic mediators is therefore of critical therapeutic importance in the development of disease and patient-specific treatment strategies.

The long term objective of this research is to explore the effects of genetic, environmental and developmental influences on the primary determinants of histamine action in atopic children and to identify potential histamine "haplotypes" that may be predictive of disease severity, progression and/or response to therapy.

The primary hypothesis is the presence of HNMT T314 allele and /or slow acetylation genotype is associated with childhood atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian, Hispanic and African American children ages 6 months to 5 years with a diagnosis of atopic dermatitis within the last 12 months will constitute the candidate pool for enrollment into the study group. The diagnosis of atopic dermatitis will be determined by the presence of at least 3 major diagnostic features (i.e., pruritis, rash,relapsing-remitting presentation, family history or atopy) in addition to at least 3 minor features (including but not limited to xerosis, elevated serum IgE, ocular involvement, food allergy). Healthy Caucasian, Hispanic and African American children within the same age range will comprise the pool for enrollment into the control group.

Exclusion Criteria:

* Any child with atopic dermatitis who has a documented history of asthma or bronchospasm or who is currently receiving treatment for either of these conditions will be excluded. Any control subject who has asthma or positive family history of allergy or atopic disease in a first-degree relative (biological mother, father or siblings) will also be ineligible for enrollment.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Caucasian,AfricanAmerican and Hispanic children with a medical diagnosis of atopic dermatitis and healthy, age matched controls
Sampling Method: Probability Sample
Enrollment: 751 (Actual)
Dates: Start 2004-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jayne Kennedy, Pharm D., Principal Investigator — Virginia Commonwealth University
Locations (7):
- United States (7):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of California at San Diego, San Diego, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - Wayne State University/Children's Hospital of Michigan, Detroit, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - Baylor College of Medicine/Texas Children's Cancer Center, Houston, Texas